CLINICAL TRIAL: NCT03034434
Title: Sonography Evaluation of Cervical Recuperation After Vaginal Delivery
Brief Title: Cervical Recuperation After Vaginal Delivery
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Other Study IDs: 0154-16-RMB
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Cervix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after vaginal delivery: Patients after vaginal delivery willing to undergo 3 trans-vaginal ultrasounds within the 48 hours after delivery.
  Interventions: Device: Trans-vaginal ultrasound

INTERVENTIONS:
Device: Trans-vaginal ultrasound — Three trans-vaginal ultrasounds, the 1st to be performed 8 hours post delivery, the 2nd 24 hours after delivery and the 3rd 48 hours after delivery.

SUMMARY:
Patients after vaginal delivery will undergo 3 trans-vaginal ultrasounds in order to examine the process of cervical recuperation post delivery.

DETAILED DESCRIPTION:
Patients after vaginal delivery will be recruited after receiving a full explanation and signing an informed consent.

The goal of the study is to examine cervical length after vaginal delivery at 3 different time intervals:

1. 8 hours post delivery.
2. 24 hours post delivery.
3. 48 hours post delivery. At each interval a trans-vaginal ultrasound will be performed, evaluating cervical length. At the end of the 3rd and final ultrasound, the patient will finish her participation in the study/ Information regarding obstetric conditions such as labor induction, gestational age at the time of delivery etc. will be collected from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Any patient after vaginal delivery.

Exclusion Criteria:

* Any patient after cesarean section.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients only.
Study Population: Patients after vaginal delivery.
Sampling Method: Non-Probability Sample
Enrollment: 1384 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cervical length after vaginal delivery. | Up to 48 hours post delivery.
  Measurement of cervical length 8, 24, 48 hours after vaginal delivery by trans-vaginal ultrasound.

SECONDARY OUTCOMES:
Differences in cervical length after vaginal delivery. | Up to 48 hours post delivery.
  Differences in cervical length after vaginal delivery as a factor of gestational age at delivery, means of labor induction, parity, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lauterbach R, Bachar G, Ben-David C, Justman N, Siegler Y, Tzur L, Copel JA, Weiner Z, Beloosesky R, Ginsberg Y. Postpartum cervical length as a predictor of subsequent preterm birth-novel insights on an old enigma. Am J Obstet Gynecol. 2023 Apr;228(4):461.e1-461.e8. doi: 10.1016/j.ajog.2022.10.012. Epub 2022 Oct 18. PMID 36265677